CLINICAL TRIAL: NCT04408443
Title: Evaluation of a Food Supplement Containing Lactobacillus Reuteri DSM 17938 + Vitamin D3 in the Prevention of Recurrent Respiratory Infections in Paediatric Patients
Brief Title: Evaluation of Lactobacillus Reuteri DSM 17938 + Vitamin D3 in the Prevention of RRI in Paediatric Patients
Acronym: LR_D3
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrollment due COVID PANDEMIA
Sponsor: Noos S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRR_D3
Record Dates: First submitted 2020-05-25; First posted 2020-05-29 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Recurrent Respiratory Tract Infections
Keywords: RRI, probiotics, vitamin D3, L. reuteri
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple (Participant, Care Provider, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reuterin D3 (Active Comparator): Patients should take 10 drops once a day during meals for 4 months followed by 2 months of follow up.
  Interventions: Dietary Supplement: Lactobacillus reuteri DSM 17938 + Vitamine D3
- Placebo (Placebo Comparator): Patients should take 10 drops once a day during meals for 4 months followed by 2 months of follow up.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri DSM 17938 + Vitamine D3 — Lactobacillus reuteri DSM 17938 (10E8 CFU in 5 drops), Vitamin D3 (400 IU in 5 drops), sunflower oil, medium chain triglycerides, silicon dioxide
  Arms: Reuterin D3
Dietary Supplement: Placebo — sunflower oil, medium chain triglycerides, silicon dioxide
  Arms: Placebo

SUMMARY:
The aim of this protocol is to evaluate, in a multicenter, randomized, double blind vs placebo clinical trial the effects of a marketed food supplement containing Lactobacillus reuteri DSM 17938 and vitamin D3 (Reuterin® D3) in the prevention of recurrent respiratory infections in pediatric patients suffered from Recurrent Respiratory Infection (RRI) in previous years.

DETAILED DESCRIPTION:
Several clinical trials documented the efficacy of probiotics in the prevention and treatment of acute gastroenteritis, while there is little evidence on the efficacy of the probiotics in the prevention of children respiratory infections.

The biological activity of probiotics is linked, partly, to their capacity to adhere to enterocytes. This would avoid the binding of pathogenic bacteria through a competitive exclusion mechanism. This inhibition toward pathogen bacteria on epithelial and mucosal level (substrate), thanks also to the production of antimicrobial substances, can have a beneficial effect on the balance of the intestinal microflora of the host and improve its immunity.

The adhesion of probiotic bacteria to the enterocyte membrane receptors influences the activation of second messengers that induces the production of cytokines. The presence of probiotic bacteria influences the commensal microorganisms in the production of lactic acid and bacteriocins. These substances inhibit the growth of pathogens and modify the balance of commensal bacteria of the intestinal bacterial flora.

Numerous controlled clinical trials show that L. reuteri DSM 17938 colonizes the human gastric and intestinal epithelium and modulates the immune response, particularly through CD4 + T-helper cells in the ileum. These data confirm the pre-clinical evidence obtained in animal models; furthermore these immunomodulatory effects may explain some clinical properties of L. reuteri DSM 17938 such as the prevention of diarrhea, inhibition of pathogen infectionand the following immune system response of the host to these pathogens, as well as the potential modulation of the immune response by the Th1/Th2 balance in the human intestinal epithelium, an answer that has been linked to the prevention and treatment of allergy. In a recent, randomized, double-blind, placebo-controlled clinical trial, L. reuteri DSM 17938, supplemented for three months to healthy children aged 6-36 months attending nursery schools, demonstrated not only a significant reduction of episodes and duration of diarrhea but also of respiratory tract infections with consequent reduction of costs for society.

Despite the prevalence of food with vitamin D and multivitamin products, reports regarding non-optimal vitamin D levels in adults and children in the world have increased, in particular among those subjects overweight and with dark pigmentation of the skin.

In addition to its well-known effects on bone health, vitamin D is indeed an important immune regulator, because it stimulates innate immunity and modulates inflammation. An analysis of data from the National Health and Nutrition Examination Survey (NHANES) between 1988 and 1994 showed an inverse relationship between vitamin D levels and the incidence of upper respiratory tract infections (URTI). These results were supported by other studies showing an increased risk of acute lower respiratory tract infections in subjects with low levels of vitamin D.

Historically, the association between rickets and the risk of serious respiratory infections is well known and vitamin D deficiency has been associated with an increased risk to contract the flu.

These considerations have led to the hypothesis that supplementation with a probiotic added with vitamin D3 may influence the composition of intestinal flora by improving the immune system and therefore reducing episodes of respiratory infections, particularly frequent during preschool age.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 1 and 6 years of age at the enrollment; both sexes
* Patients with an history of RRI, according to the definition (The definition of Recurrent respiratory infections (RRI) is the onset of 8 or more documented airway infections during the year, in preschool children (up to three years of age) or 6 or more in children older 3 years, in the absence of any other underlying pathological condition) in the previous year.
* Atopic and non-atopic patients
* Willing and able to give informed consent of participation in the study by parent or legal guardian.

Exclusion Criteria:

* Presence of autoimmune diseases, immunodeficiency, neuromuscular diseases, congenital cardiomyopathies, metabolic diseases
* Patients in therapy with other drugs for the treatment of RRI
* Supplementation with probiotics and /or prebiotics in the previous 2 weeks
* Vitamin D intake in the last 4 weeks
* IgA deficiency
* Antibiotic treatment at least 4 week before in inclusion
* Participation in other clinical trials

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change of the number of respiratory infection | 4 months + 2 months of follow up
  Change of the number of respiratory infection respect the previous year

SECONDARY OUTCOMES:
Change of number of days with fever | 4 months + 2 months of follow up
  To evaluate the change of the number of days with fever
Change of the antibiotic use | 4 months + 2 months of follow up
  To evaluate the change of the antibiotic use
Change of number of visit to Pediatrician | 4 months + 2 months of follow up
  To evaluate the change of the number of visit to Pediatrician
Change of number of days of absence from the nursery / kindergarten | 4 months + 2 months of follow up
  To evaluate the change of the number of days of absence from the nursery / kindergarten
Changes of days of absence from work by parents | 4 months + 2 months of follow up
  To evaluate the change of days of absence from work by parents
Modification of intestinal microflora | 4 months + 2 months of follow up
  To evaluate the modification of intestinal microflora

CONTACTS AND LOCATIONS:
Overall Officials: Michele Miraglia del Giudice, Prof., Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- University of Campania Luigi Vanvitelli, Naples, Italy

IPD SHARING:
Plan to Share IPD: No